CLINICAL TRIAL: NCT07304856
Title: Prospective Observational Study of the Role of Extracellular Vesicles (EVs) as Biomarkers of Pulmonary Involvement in Patients With Sporadic Lymphangioleiomyomatosis (S-LAM) and Tuberous Sclerosis Complex-Associated LAM (TSC-LAM)
Brief Title: Role of Extracellular Vesicles as Biomarkers of Pulmonary Involvement in Patients With Lymphangioleiomyomatosis and Tuberous Sclerosis Complex
Status: Recruiting | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Michele Mondoni, MD, associated professor of respiratory medicine, University of Milan
Other Study IDs: LAM_EVs
Record Dates: First submitted 2025-09-15; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-09

CONDITIONS: Lymphangioleiomyomatosis (LAM); Extracellular Vesicles; Generation and Function
Keywords: LAM, TSC, EVs
MeSH Terms: conditions — Lymphangioleiomyomatosis | interventions — Respiratory Function Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- S-LAM: Patients with sporadic LAM
  Interventions: Diagnostic Test: Pulmonary Function Test; Diagnostic Test: Analysis of Extracellular Vesicles
- TSC-LAM: Patients with TSC-associated LAM
  Interventions: Diagnostic Test: Pulmonary Function Test; Diagnostic Test: Analysis of Extracellular Vesicles
- TSC: Patients with TSC and no pulmonary involvement
  Interventions: Diagnostic Test: Pulmonary Function Test; Diagnostic Test: Analysis of Extracellular Vesicles
- Control: Healthy subjects
  Interventions: Diagnostic Test: Pulmonary Function Test; Diagnostic Test: Analysis of Extracellular Vesicles

INTERVENTIONS:
Diagnostic Test: Pulmonary Function Test — Spirometry, Plethysmography, Diffusing capacity of the lungs for carbon monoxide (DLCO), and Six-minute walk test (6MWT).
Diagnostic Test: Analysis of Extracellular Vesicles — From the venous blood sample, plasma will be separated, and extracellular vesicles (EVs) will be isolated through serial centrifugation steps. The EVs will be analyzed to assess their concentration (particles/mL) and size (nanometers, nm). Additionally, omics analyses will be performed to study the molecular content of the EVs, including nucleic acids, proteins, and lipids.

SUMMARY:
Lymphangioleiomyomatosis (LAM) is a rare lung disease, linked to Tuberous Sclerosis Complex (TSC) or occurring sporadically, and involves abnormal mTORC1 activation. LAM cells are neoplastic, and recent focus has turned to extracellular vesicles (EVs), which mediate tumor progression and may serve as biomarkers. This study, conducted at the Pulmonology Unit of ASST Santi Paolo e Carlo and the Pharmacology Laboratory of the University of Milan, will analyze the characteristics of serum EVs in patients with LAM and TSC. During scheduled outpatient visits, clinical and functional data and blood samples will be collected. Plasma will be separated, and EVs will be isolated via centrifugation. EVs will be analyzed for size, concentration, and molecular content (proteins, lipids, nucleic acids). The results obtained will be collected and correlated with the clinical and functional data.

ELIGIBILITY:
Inclusion Criteria:

Female participants aged ≥18 years Confirmed diagnosis of tuberous sclerosis complex (TSC) and/or lymphangioleiomyomatosis (definite diagnosis of TSC-LAM or S-LAM) Follow-up at the Pulmonology Unit of ASST Santi Paolo e Carlo, Milan Ability to provide written informed consent

Exclusion Criteria:

Diagnosis of "probable" or "possible" LAM Refusal to provide written informed consent

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female participants aged ≥18 years with a confirmed diagnosis of tuberous sclerosis complex (TSC) and/or lymphangioleiomyomatosis (LAM), followed at the Pulmonology Unit of ASST Santi Paolo e Carlo, Milan, and able to provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2026-01-16 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
To compare the number and morphological characteristics of Extracellular Vesicles (EVs) in women with S-LAM, TSC-LAM, TSC without pulmonary involvement, and healthy controls | One year
  The concentration (particles/mL) and the size (nm) of EVs isolated from the plasma of 3 groups of patients (sporadic LAM, LAM associated to TSC, TSC without pulmonary involvement) and of 1 healthy control group will be assessed through Nanoparticle Tracking Analysis.

SECONDARY OUTCOMES:
To evaluate the content of EVs (miRNA, lipids, proteins, metabolites) through omics analyses in women with S-LAM, TSC-LAM, TSC without pulmonary involvement, and healthy controls | One year
  The content of EVs isolated from the plasma of 3 groups of patients (plasma of 3 groups of patients (sporadic LAM, LAM associated to TSC, TSC without pulmonary involvement) and of 1 healthy control group will be assessed through
  -omics analyses.
Effect of mTOR-inhibitor therapy on EVs count | One year
  The concentration (particles/mL) of extracellular vesicles (EVs) in patients with LAM treated with mTOR inhibitor therapy (sirolimus or everolimus) compared with patients not receiving mTOR inhibitor therapy will be assessed using Nanoparticle Tracking Analysis (NTA).
Effect of mTOR-inhibitor therapy on EVs morphology | One Year
  The size (nanometers, nm) of extracellular vesicles (EVs) in patients with LAM treated with mTOR inhibitor therapy (sirolimus or everolimus) compared with patients not receiving mTOR inhibitor therapy will be assessed using Electron Microscopy (EM).
Association between EVs characteristics and disease severity | One year
  The concentration (particles/mL) and size (nanometers, nm) of extracellular vesicles (EVs) isolated from the plasma of patients with S-LAM, TSC-LAM, and TSC without pulmonary involvement will be analyzed for their association with disease severity, as assessed by the number of systemic manifestations of TSC and the presence of pulmonary disease.
Association between EVs characteristics and pulmonary disease severity | One year
  The concentration (particles/mL) and size (nanometers, nm) of extracellular vesicles (EVs) isolated from the plasma of patients with LAM (including both S-LAM and TSC-LAM) will be analyzed for their association with disease severity, based on the number of pulmonary complications, including pneumothoraces, chylothoraces, development of respiratory failure, and the need for lung transplantation.
Association between EVs characteristics and pulmonary function | One year
  The concentration (particles/mL) and size (nanometers, nm) of extracellular vesicles (EVs) isolated from the plasma of patients with LAM (including both S-LAM and TSC-LAM) will be analyzed for their association with pulmonary function, as measured by spirometry and diffusion parameters (FEV1, FVC, and DLCO), with FEV1 and FVC expressed in liters and % predicted, and DLCO expressed as % predicted.

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonology Unit ASST Santi Paolo e Carlo, Ospedale San Paolo, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided